CLINICAL TRIAL: NCT02164552
Title: Vitamin D Status in Relation to Insulin Sensitivity, Resistance and Inflammatory Response Among Saudi Women With Polycystic Ovary Syndrome
Brief Title: Vitamin D Status in Relation to Insulin Sensitivity Among Saudi Women With Polycystic Ovary Syndrome
Acronym: CEOR-04-08
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mohammed-Salleh M. Ardawi, Professor, King Abdulaziz University
Other Study IDs: CEOR-04-08; Vitamin D PCOS (Other Grant/Funding Number: CEOR/001-08 and CEOR/004-08)
Record Dates: First submitted 2014-06-10; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; vitamin D; insulin resistance; glycemic control
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Vitamin D3 pills: Vitamin D3 (cholecalciferol) supplementation (50,000 IU/week for 8 weeks) followed by 1000 IU/day for 16 weeks
  Interventions: Dietary Supplement: Vitamin D3 pills
- Placebo pill: Placebo pills will be given 1 per week for 8 weeks followed by 1 per day for 16 weeks
  Interventions: Other: Placebo pills

INTERVENTIONS:
Dietary Supplement: Vitamin D3 pills — Dietary supplement
  Other Names: Vitamin D3; (cholecalciferol)
  Groups: Vitamin D3 pills
Other: Placebo pills — Placebo pills similar in appearance and shape but without vitamin D
  Groups: Placebo pill

SUMMARY:
The study tests the hypothesis that correction of vitamin D deficiency among women with PCOS will improve insulin sensitivity and resistance and inflammatory response to PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common complex and heterogenous endocrine disorder. It affects ≤10% of women of reproductive age, with approximately 16%-80% of the affected women being obese. Polycystic ovary syndrome frequently is associated with insulin resistance (IR) accompanied by compensatory hyperinsulinemia, and IR is aggravated by the interaction between obesity and the syndrome. Moreover, the contribution of body mass and/or body fat distribution to IR of PCOS remains controversial. In addition, women with PCOS with IR are at an increased risk of developing diabetes, hypertension, dyslipidemia and atherosclerosis. Preliminary data on the local women with PCOS showed high prevalence of vitamin D deficiency (serum 25(OH)D < 50 nmol/L). Recent studies showed that vitamin D deficiency is linked to IR, type 2 diabetes mellitus, obesity, inflammation and cardio vascular disease. Several studies have demonstrated that serum 25(OH)D levels were negatively correlated with body mass index (BMI), body fat, and IR. These conditions are common among women with PCOS. Accordingly, it is anticipated that vitamin D deficiency and/or insufficiency may contribute to the endocrine and metabolic disarrangements among women with PCOS. Such adverse effects may further contribute to the risk of further long term complications among women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

PCOS diagnosis to include three of the Rotterdam criteria

Exclusion Criteria:

pregnancy lactation taking vitamin d or calcium supplement in excess of a regular multivitamins diabetes mellitus uncontrolled hypertension liver disease renal disease secondary causes of hyperandrogenism metabolic bone disease thyroid dysfunction taking oral contraceptives taking hypoglycemic agents (metformin or thiazolidinediones) medication to affect plasma sex steroids for >/3 months before the study smokers

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women were recruited through Infertility clinics at King Abdulaziz University Hospital, New Jeddah Clinic Hospital and Dr S Fakeeh Hospital, Jeddah area during general health survey and consecutively referred to a special clinic at the Center of Excellence for Osteoporosis Research for enrollment at the present study
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Correction of vitamin D deficiency improves insulin resistance compared to placebo | 24 weeks
  The primary endpoint was an improvement in insulin resistance parameters [Fasting serum insulin,glucose-to-insulin ratio (GIR) and homeostasis model assessment (HOMA) ] from baseline and at 24 weeks in vitamin D supplemented as compared with placebo groups.

SECONDARY OUTCOMES:
Insulin sensitivity | 24 weeks
  Secondary endpoints were changes in parameter of insulin sensitivity[ quantitative insulin sensitivity check index (QUICKI)], among vitamin D supplemented group vs placebo group from baseline and at the end of the trial

OTHER OUTCOMES:
Exploratory and safety outcome | 24 weeks
  Other endpoints were changes in inflammatory markers (hs-CRP)
Exploratory outcomes: lipid profile | 24 weeks
  Other endpoints were changes in lipid profile (total cholesterol, HDL-c, LDL-c, and triglycerides)
Exploratory outcomes: liver and renal function tests | 24 weeks
  Other endpoints were changes in liver function tests [albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase(ALP)]; renal function tests (cystatine C, uric acid, urea) and parathyroid hormone (PTH)
Exploratory outcomes: glycemic control | 24 weeks
  Other endpoints were changes in HbA1c, fasting plasma glucose and fasting plasma insulin
Exploratory outcomes: vitamin D status | 24 weeks
  Other endpoints were changes in serum 25-hydroxyvitamin D
Exploratory outcomes: endocrine profile | 24 weeks
  Other endpoints were changes in (follicle-stimulating hormone, luteinizing hormone, prolactin, thyroid-stimulating hormone, free thyroxine, total testosterone, dehydroepiandrosterone (DHEA), DHEA sulfate, delta 4-androstenedione and sex-hormone binding globulin).

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahim A Rouzi, FRCPC, Principal Investigator — Center of Excellence for Osteoporosis Research and Faculty of Medicine, King Abdulaziz University; Mohammed-Salleh M Ardawi, PhD, FRCPath, Study Director — Center of Excellence for Osteoporosis Research, and Faculty of Medicine, King Abdulaziz University
Locations (1):
- Center of Excellence for Osteoporosis Research, King Abdulaziz University, Jeddah, Mecca Region, Saudi Arabia